CLINICAL TRIAL: NCT02338869
Title: Psycho-Social Well Being Following Stroke - A Randomized Controlled Trial
Brief Title: Psycho-Social Well Being Following Stroke
Acronym: PsychoStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Marit Kirkevold, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/2047
Record Dates: First submitted 2014-10-04; First posted 2015-01-14 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialogue-based psychosocial intervention (Experimental): Participants receive six individual meetings with trained health care professional in additional to usual rehabilitation and care. Dialogues focus on individual psychosocial challenges and needs and provide emotional and informational support to encourage and facilitate coping.
  Interventions: Behavioral: Dialogue-based psychosocial rehabilitation
- Usual care Control group (No Intervention): Participants receive usual rehabilitation and care.

INTERVENTIONS:
Behavioral: Dialogue-based psychosocial rehabilitation
  Arms: Dialogue-based psychosocial intervention

SUMMARY:
Multicenter randomized controlled trial (RCT) testing the effect of a dialogue-based psychosocial intervention for stroke acute survivors in primary care one to six months poststroke. Primary outcome is psycho-social health and wellbeing, measured by GHQ28 (primary outcome) and SAQoL (secondary outcome). 400 stroke survivors are randomized into intervention group or control group. Patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* being adults (over 18 years old),
* suffered an acute stroke within the last month,
* medically stable,
* sufficient cognitive functioning to participate (assessed by their physician/stroke team and acceptable Raven's score (see below),
* interested in participating,
* able to understand and speak Norwegian, and
* able to give informed consent.

Exclusion Criteria:

* moderate to severe dementia or other serious disease.

Persons with aphasia will be examined by a speech therapist and excluded if they have significant impressive aphasia or severe expressive aphasia inconsistent with participating in the dialogues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire (GHQ 28) | T2 (6 months poststroke)
  28 item general scale measuring emotional distress. Four subscales (somatic symptoms, anxiety/insomnia, social dysfunction and serious depression

SECONDARY OUTCOMES:
The Stroke and Aphasia Quality of Life scale (SAQOL-39) | T2 (6 months poststroke)
  Disease-specific quality of life scale, measures patient's perspective of stroke's impact on 'physical', 'psychosocial' and 'communication' domains.

CONTACTS AND LOCATIONS:
Overall Officials: Marit Kirkevold, Ed.D, Principal Investigator — University of Oslo
Locations (1):
- Oslo University hospital, Oslo, Norway

REFERENCES:
- [Derived] Mangset M, Kitzmuller G, Evju AS, Angel S, Aadal L, Martinsen R, Bronken BA, Kvigne KJ, Bragstad LK, Hjelle EG, Sveen U, Kirkevold M. Perceived study-induced influence on the control group in a randomized controlled trial evaluating a complex intervention to promote psychosocial well-being after stroke: a process evaluation. Trials. 2021 Nov 27;22(1):850. doi: 10.1186/s13063-021-05765-w. PMID 34838094
- [Derived] Martinsen R, Kitzmuller G, Mangset M, Kvigne K, Evju AS, Bronken BA, Bragstad LK, Hjelle EG, Sveen U, Kirkevold M. Nurses' and occupational therapists' experiences of conducting a home-based psychosocial intervention following stroke: a qualitative process evaluation. BMC Health Serv Res. 2021 Aug 11;21(1):791. doi: 10.1186/s12913-021-06857-8. PMID 34376188
- [Derived] Bragstad LK, Lerdal A, Gay CL, Kirkevold M, Lee KA, Lindberg MF, Skogestad IJ, Hjelle EG, Sveen U, Kottorp A. Psychometric properties of a short version of Lee Fatigue Scale used as a generic PROM in persons with stroke or osteoarthritis: assessment using a Rasch analysis approach. Health Qual Life Outcomes. 2020 Jun 5;18(1):168. doi: 10.1186/s12955-020-01419-8. PMID 32503548
- [Derived] Hjelle EG, Bragstad LK, Zucknick M, Kirkevold M, Thommessen B, Sveen U. The General Health Questionnaire-28 (GHQ-28) as an outcome measurement in a randomized controlled trial in a Norwegian stroke population. BMC Psychol. 2019 Mar 22;7(1):18. doi: 10.1186/s40359-019-0293-0. PMID 30902115
- [Derived] Bragstad LK, Bronken BA, Sveen U, Hjelle EG, Kitzmuller G, Martinsen R, Kvigne KJ, Mangset M, Kirkevold M. Implementation fidelity in a complex intervention promoting psychosocial well-being following stroke: an explanatory sequential mixed methods study. BMC Med Res Methodol. 2019 Mar 15;19(1):59. doi: 10.1186/s12874-019-0694-z. PMID 30876403
- [Derived] Kirkevold M, Kildal Bragstad L, Bronken BA, Kvigne K, Martinsen R, Gabrielsen Hjelle E, Kitzmuller G, Mangset M, Angel S, Aadal L, Eriksen S, Wyller TB, Sveen U. Promoting psychosocial well-being following stroke: study protocol for a randomized, controlled trial. BMC Psychol. 2018 Apr 3;6(1):12. doi: 10.1186/s40359-018-0223-6. PMID 29615136